CLINICAL TRIAL: NCT02188459
Title: Placebo-controlled Trial of Bupropion for Smoking Cessation in Pregnant Women
Acronym: BIBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Kranzler (Other)
Responsible Party: Sponsor-Investigator, Henry Kranzler, M.D., University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 820364
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupropion (Active Comparator): Bupropion 150 mg BID, PO for 10 weeks
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Placebo BID, PO for 10 weeks. The formulation appears identical to the bupropion capsules.
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — A total of 360 participants will be randomly assigned to one of two treatment conditions: Bupropion 300 mg/day (n = 180) or placebo (n = 180). We will use small-block randomization by site (Penn). A PHQ-9 score of 10 or greater will be used to identify major depression and stratify the randomization on it. Study site (Penn) will be the second of the two stratification variables.
  Other Names: Wellbutrin

SUMMARY:
Smoking during pregnancy adversely affects the health of the mother and her developing baby. Maternal smoking approximately doubles the risk of miscarriage, placental complications, preterm delivery, low birth weight and fetal and newborn death. The most common adverse effect of smoking during pregnancy is low birth weight, which sharply increases the risk of the newborn becoming ill or dying. In the US, maternal smoking is responsible for 30% of low birth weight babies, 10% of premature deliveries, and 5% of infant deaths. Fortunately, smoking cessation by pregnancy week 16, or as late as the third trimester, results in a near-normal weight infant at birth. Even reductions in smoking increase birth weight.

Despite the known risks, the majority of women who are smoking at the time of their first prenatal visit continue to smoke. Bupropion is approved by the US Food and Drug Administration (FDA) for smoking cessation in people who are not pregnant, but there are no carefully controlled studies on the use of Bupropion to help pregnant women quit smoking. Bupropion is also FDA approved to treat depression, and some pregnant women have taken it for that purpose, even though it has not been formally tested. The investigators propose to conduct a randomized, parallel-group, double-blinded, placebo-controlled, 10 week trial of Bupropion in 360 pregnant women who smoke daily and wish to quit smoking.

The study has three primary hypotheses. First, the investigators hypothesize that Bupropion treated subjects will decrease the frequency of smoking more than placebo-treated subjects. Second the investigators hypothesize that Bupropion treated subjects will have greater positive pregnancy and child health outcomes than placebo-treated subjects. Third the investigators hypothesize that Bupropion treated subjects will have decreased frequency of depressive symptoms and cigarette craving than placebo-treated subjects. These finding will provide information on the safety and efficacy of bupropion treat for smoking cessation in pregnant women.

DETAILED DESCRIPTION:
A. General Design: This is a phase II, prospective, placebo-controlled randomized controlled trial of the efficacy and safety of bupropion in combination with behavioral counseling for smoking cessation during pregnancy. Pregnant smokers (N=360) will receive bupropion or placebo treatment for 10 weeks, under strict double-blind conditions, with 3 post-treatment follow-up sessions: 2 and 6 weeks postpartum (with counseling to prevent relapse or encourage a repeat quit attempt) and monitoring of the persistence of treatment effects at 24 weeks post-quit date.

B. Recruitment: We will distribute IRB (Institutional Review Board)-approved brochures and posters to recruit pregnant women who smoke and wish to quit smoking through participation in the trial. At Penn Medicine sites, we will access the hospitals' EPIC computer programs to identify pregnant smokers receiving prenatal care and, working with their obstetrician, invite them to consider study participation. We will conduct a brief screening interview over the phone or in-person at the participant's obstetrics clinic to assess study eligibility criteria. Prospective participants who appear to meet eligibility criteria for the study will be scheduled for an in-person Informed Consent and Screening visit.

C. Screening Visit: Participants will read and sign the informed consent form, after all of their questions have been answered. Participants will then be asked to provide the researchers with information to determine whether they are eligible to participate in the study. On this visit, participants will be interviewed for about an hour. This interview will include questions about medical and pregnancy history, and any mood or other symptoms and determine the baby's date of delivery. We will also ask about any past or current use of alcohol, drugs, and cigarettes.

D: Baseline Visit: This in-person visit will be completed within 30 days of the screening visit and will last approximately 90 minutes. At the visit, we will measure heart rate and complete questionnaires by telephone and in person. We will take a blood sample (3 tubes, enough to fill 1.5 tablespoons) to be used to conduct genetic testing and to measure the body's ability to break down nicotine, which is contained in cigarettes.

At this visit participants will receive the first of six counseling sessions in the study. This first, "pre-quit" counseling session will last 30 minutes and will help to prepare them to quit smoking. They will be given study medication at this visit and will be instructed to begin taking it the following morning. They will be asked to identify a quit date within a week of beginning the study medication. They will start the study medication by taking one capsule (150 mg/day or placebo, a harmless, inactive substance) each morning for the first 3 days and then one capsule each morning and each evening (150 mg twice daily) for the remainder of the 10-week study treatment period. At this visit, and at every visit while taking the study medication, we will record any side effects that may have been experienced from the study medication. We will also ask participants to return all study medication that they have not taken and the study medication bottle.

The day after the Baseline Visit, the participants will begin to receive two daily text messages. The first message of the day (in the morning) will provide information on the expected development based on the baby's age, accompanied by a reminder to take the study medication. The second message of the day (in the evening) will ask the participants whether they took all of their study medication that day. They'll be asked to text back indicating that they received the message (in the morning) and whether they took the medication that day (in the evening). We will ask them which times they would like to receive the text messages each day. Although the information that they provide will help us to keep track of their participation, the inbox for our texting center is not monitored, so we will direct them to call our study staff to speak with them directly, rather than texting them if they have any study-related questions.

Visit C: Quit Date Visit: The scheduled quit date visit will occur approximately one week after the baseline visit and will last approximately 45 minutes. During this visit, we will measure the participants' heart rate and ask them to blow into an instrument that measures a chemical (carbon monoxide) that is in tobacco smoke. The study nurse will collect any medication not taken and the study medication bottle. The participants will receive a four-week supply of study medication and a study nurse will ask them about any study medication side effects that they may have experienced since starting the study. They will also be asked to complete some questionnaires and will receive 20 minutes of "quit-day" counseling, which will help them to identify things that could cause them to return to smoking and to develop a plan to avoid tempting situations.

Visit D: Week 3: This visit will occur by telephone and will last approximately 25 minutes, during which time the participants will be asked to complete questionnaires over the telephone. They will be asked about their cigarette use since the last visit and any medication side effects they may have experienced. They will also receive 10 minutes of counseling by phone to help them avoid smoking or, if they need to, set another quit date to try again to quit smoking.

Visit E: Week 5: This in-person visit will last approximately 30 minutes. The participants will be asked to complete some questionnaires and be interviewed about their cigarette use since the last visit. We will measure their heart rate and they will be asked to blow into an instrument that measures a chemical (carbon monoxide) that is in tobacco smoke. They will be asked to provide a blood sample (2 tubes, enough to fill 1 tablespoon) to be used to measure the concentration of study medication in the blood. The study nurse will collect any medication that the participants have left as well as the study medication bottle. They will receive a five-week supply of study medication and a study nurse will ask them about any study medication side effects that they may have experienced since starting the study. They will also receive 10 minutes of counseling to help they avoid smoking or, if needed, set another quit date to try quitting again.

Visit F: Week 7: This telephone visit will last approximately 15 minutes. The participants will be asked to complete some questionnaires. They will also be asked about their cigarette use since the last visit and any medication side effects they may have experienced.

Visit G: Endpoint visit: This in-person visit will last approximately 25 minutes. The participants will be asked to complete questionnaires and about their cigarette use since the last visit. During the visit we will measure their heart rate and they will be asked to blow into an instrument that measures a chemical (carbon monoxide) that is in tobacco smoke. The study nurse will collect any medication that they had not taken and the study medication bottle. The study nurse will ask them about any study medication side effects that they may have experienced since starting the study.

Visit H: Week 24 after the Quit Date: About six months after the participants started treatment, they will be contacted by telephone. During this phone call, a research technician will complete several questionnaires with them, similar to those they completed previously. Some participants will be asked to come back to the center following this interview to provide carbon monoxide breath samples as they did previously. Approximately two weeks prior to the phone call we may send a reminder letter that the phone visit is coming up.

Visits I and J: 2 and 6 weeks after delivery: The last two sessions will be held by telephone after the birth of the baby. The participants will be asked to complete several questionnaires, similar to those completed previously. They will also receive 10 minutes of counseling over the phone.

ELIGIBILITY:
Inclusion Criteria:

1. Currently smoking on average 3 or more cigarettes per day for the preceding 7 days with a breath CO of at least 5 ppm and wants to quit smoking
2. Pregnant at 13-26 weeks gestation (to maximize safety and the likelihood of receiving 10 weeks of treatment)
3. >18 years of age
4. Able to speak and read English at a 6th grade level or higher, using the Slosson Oral Reading Test (SORT)
5. Committed to remaining in the geographic area for at least 3 months postpartum
6. Able to sign written informed consent and commit to completing the procedures involved in the study.
7. Methadone or buprenorphine-maintained women must be in methadone or buprenorphine treatment for a minimum of 2 weeks prior to entering the study. Their 2 most recent urine drug screens, consecutive and administered at least one week apart, must both be positive for methadone or buprenorphine and negative for drugs of abuse other than cannabis. Participants who screen positive for other drugs at either time point will not be enrolled in the study until they meet this criterion.

Exclusion Criteria:

1. During the last 90 days from screening visit, meets any criteria for a DSM-IV diagnosis of drug or alcohol dependence-excluding tobacco or cannabis dependence and, for methadone or buprenorphine maintenance patients, opioid dependence-AND either evidences ongoing use of illicit drugs other than cannabis or continues to abuse or misuse prescription drugs such as CNS stimulants.
2. Pregnant with triplets or higher order multiple gestations
3. Has an unstable psychiatric disorder (i.e., suicide risk moderate or severe, as reflected by a score of >9 on the MINI Section B (Suicidality) or a suicide attempt during the preceding year, psychiatric hospitalization within the last 3 months; current psychotic disorder based on the MINI)
4. Current or past Bipolar Disorder as determined by a study psychiatrist or psychologist based on assessment with the MINI, relevant information from the medical record and, when warranted, direct clinical evaluation.
5. Current, regular use of psychotropic medication, inhibitors of CYP2B6 (e.g., ticlopidine, clopidogrel), inducers of CYP2B6 (e.g., ritonavir, lopinavir, efavirenz), anticonvulsants (e.g., carbamazepine, phenobarbital, phenytoin), beta-blockers (e.g., metoprolol), Type 1C antiarrhythmics (e.g., propafenone and flecainide), drugs that require metabolic activation by CYP2D6 to be effective (e.g., tamoxifen), drugs that lower seizure threshold (e.g., antipsychotics, tricyclic antidepressants, theophylline, or systemic corticosteroids), levodopa or amantadine
6. Current unstable medical problems or potential inability to tolerate study treatment [e.g., threatened abortion: current persistent hyperemesis gravidarum (HEG) requiring intravenous fluids (to be rescreened when HEG is stabilized/resolved and no electrolyte abnormalities are evident); hypertension with evidence of end organ dysfunction or on more than 2 medications at the start of the pregnancy]; arteriovenous malformation; AIDS; laboratory evidence of hepatic impairment (e.g. viral hepatitis with serum transaminase levels more than twice the upper limit of normal) ; renal impairment (e.g., elevated creatinine or creatinine clearance <75cc/hr), metabolic disorders (e.g., hypoglycemia, hyponatremia) or end organ damage from any chronic medical condition (e.g. abnormal pulmonary function tests), glaucoma, or other significant medical problems that in the opinion of a study obstetrician makes the risk of study participation unacceptable.
7. Known major fetal congenital malformation-as determined by the study obstetrician-diagnosed prior to study randomization
8. History of seizure disorder
9. Current use of a smoking cessation medication in addition to the study medication, such as nicotine replacement therapy
10. Current or history of bulimia or anorexia nervosa
11. Current use of tobacco products other than cigarettes (e.g., E-cigarettes)
12. Current clinically significantly abnormal laboratory evaluations that are not adequately controlled by standard of care treatment.
13. History of severe head injury (i.e., with loss of consciousness)
14. Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigator and/or Study Physician.
15. Inability to provide informed consent or judged by the Principal Investigator and/or Study Physician to be an unsuitable candidate for a clinical drug trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Kranzler, M.D., Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Christiana Care Health System, Newark, Delaware
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kranzler HR, Washio Y, Zindel LR, Wileyto EP, Srinivas S, Hand DJ, Hoffman M, Oncken C, Schnoll RA. Placebo-controlled trial of bupropion for smoking cessation in pregnant women. Am J Obstet Gynecol MFM. 2021 Nov;3(6):100315. doi: 10.1016/j.ajogmf.2021.100315. Epub 2021 Jan 22. PMID 33493703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of pregnant smokers began on 10/30/2014. The study completed all treatment and follow-up phases on 1/20/2020. Pregnant smokers were recruited from maternal medicine sites in Philadelphia, PA and Newark, DE.
Period: Overall Study
Arm/Group | Bupropion | Placebo
Started | 64 | 65
Completed | 61 | 58
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 4
Not completed — Early Termination | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo BID, PO for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Bupropion | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (4.7) | 29.0 (5.0) | 28.5 (4.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 32 | 67
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 64 | 129
Education (% High School Graduate or less) [Count of Participants; unit: Participants] | 21 | 18 | 39
Annual Household Income (<40K) [Count of Participants; unit: Participants] | 49 | 47 | 96
Marital Status (% Partnered) [Count of Participants; unit: Participants] | 25 | 22 | 47
Depression (PHQ-9) [Mean (Standard Deviation); unit: Total score] — The Patient Health Questionnaire (PHQ-9), is a validated 9-item self-report measure of depressive symptoms that yields a total score of 0-27 (Kroenke, Spitzer et al. 2001). A PHQ-9 score of 10 or greater was used to identify major depression. The higher the score the great the symptoms of depression.
  Total score | 4.9 (3.8) | 5.4 (4.1) | 5.1 (3.9)
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: Total score] — Fagerstrom Test for Nicotine Dependence (FTND) (Fagerstrom and Schneider 1989) is a 6-item, self-report measure of nicotine dependence derived from the Fagerstrom Tolerance Questionnaire.
  The range is from 1-8 with a higher score indicating a greater level of nicotine dependence.
  Total score | 3.8 (1.9) | 3.8 (1.9) | 3.8 (1.9)
Cigarettes/Day in Past 30 Days [Mean (Standard Deviation); unit: Cigarettes per day] — Number of cigarettes smoke each day over the past 30 days was collected using the Timeline Follow-back method, combined with the exhaled carbon monoxide (CO) concentrations. Abstinence was self-reported and confirmed by a CO concentration <8 parts per million (ppm). A CO of 8 ppm or greater indicates cigarettes smoked where smoked with higher CO ppm concentration indicates that a greater number of cigarettes were smoked. Participants were assumed to be smoking if they did not provide self-report data or a breath sample at the time of measurement.
  Cigarettes per day | 7.9 (4.5) | 8.0 (4.2) | 7.9 (4.3)
Breath CO, ppm [Mean (Standard Deviation); unit: parts per million] — Breath Carbon Monoxide (CO) is measured in parts per million (ppm) using a hand held breath CO analyzing device. The device measures CO in a range from 0 ppm to 25 ppm, 25 ppm being the greatest concentration of CO the device can measure. Self reported abstinence was confirmed by a breath CO concentration <8 ppm.
  parts per million | 8.3 (5.2) | 9.2 (5.7) | 8.8 (5.4)
Total number of years smoking cigarettes [Mean (Standard Deviation); unit: Totals years smoking cigarettes] — Participants responded to a questionnaire that queried the total number of years that they had been smoking cigarettes. More years of smoking is associated with greater severity of nicotine dependence and greater difficulty in quitting smoking.
  Totals years smoking cigarettes | 12.0 (5.5) | 13.0 (5.1) | 12.5 (5.3)
Number of Times Quit Smoking for >24 Hours [Mean (Standard Deviation); unit: number of times quit smoking cigarettes] — Participants responded to a question regarding the total number of times that they quit smoking cigarettes for a period greater than 24 hours.
  number of times quit smoking cigarettes | 2.9 (2.7) | 3.8 (7.0) | 3.3 (5.3)
Weeks of Gestational Age [Median (Standard Deviation); unit: Weeks] — Gestational Age is measured in weeks. Only pregnant smokers who had a gestational age between 13 and 26 weeks were included in the study. Gestational age was assessed usin a method developed by the NICHD-sponsored Maternal-Fetal Medicine Units Network. The gestational age was based on the projected estimated date of delivery (EDD), as determined by ultrasound (U/S) and the last menstrual period (LMP).
  Weeks | 18.5 (4.6) | 18.4 (4.2) | 18.4 (4.4)
Number of Pregnancies [Mean (Standard Deviation); unit: pregnancies] — Number of pregnancies was reported by the patient in response to a query and confirmed with medical record review when available.
  pregnancies | 3.5 (1.9) | 4.2 (2.6) | 3.8 (2.3)
History of Premature Delivery [Count of Participants; unit: Participants] | 11 | 14 | 25
History of Ectopic Pregnancy [Count of Participants; unit: Participants] | 2 | 4 | 6
History of Miscarriage [Count of Participants; unit: Participants] | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cessation Success at Week 10 After Target Quit Date
Description: Participants will be considered to be abstinent if they self-report abstinence (not even a puff of a cigarette) for >7 days prior to the assessment after 10 weeks of treatment post-To Quit Day and have a CO <8 ppm at that time. As per convention, participants are assumed to be smoking if they self-report to be smoking at the time point, cannot be reached to provide data at the time point, fail to provide a breath sample at the time point, or provide a breath sample at the time point that has a CO concentration >8 ppm.
Time Frame: 10 weeks
Population: We tested treatment group differences as a binary abstinence outcome using a repeated measure generalized estimating equations (GEE) model with a logit link. Point prevalence quit rates at the end of week 10 of treatment post-TQD were the primary outcome variables.
Measure: Number; unit: Participants with cessation success
Groups:
- Placebo Group: 10 mg placebo daily 10 weeks
- Bupropion Group: 10 mg buproprion 10 weeks
Arm/Group | Placebo Group | Bupropion Group
Number analyzed (Participants) | 65 | 64
Participants with cessation success | 12 | 7

2. Primary Outcome: Number Moderate or Severe Side Effects
Description: For adverse effects, our primary outcome will be the frequency of moderate or severe side effects from a checklist of bupropion-related side effects (derived from completed bupropion studies), as well as those elicited with open-ended questions, through regular obstetrics visits, and assessments triggered by any pregnancy-related complication. Adverse effects will be systematically assessed by study personnel at 5 time points over the course of the 10-week study and can trigger dose reductions or suspension of medication.
Time Frame: 10 week treatment phase
Measure: Mean (Standard Deviation); unit: adverse effects
Arm/Group | Placebo | Bupropion
Number analyzed (Participants) | 65 | 64
adverse effects | .7 (1.2) | 1.1 (1.8)

3. Primary Outcome: Birth Outcomes for Gestational Age
Description: Birth outcomes obtained from labor and delivery records gestational age, measured in weeks.
Time Frame: Postpartum
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 64 | 65
weeks | 37.1 (4.7) | 38.1 (1.7)

4. Primary Outcome: Birth Weight Outcomes
Description: Birth weight outcomes were obtained from labor and delivery clinical records. Birth weight is measure in grams.
Time Frame: Postpartum
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 64 | 65
grams | 2925.9 (680.5) | 2996.5 (521.7)

5. Primary Outcome: Birth Outcomes, Size (Percentile) for Gestational Age.
Description: Birth outcomes obtained from labor and delivery records infant size for gestational age, whether small for gestational age (i.e., <10th percentile birth weight for gestational age as determined by the Alexander curve).
Time Frame: Postpartum
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 64 | 65
percentile | 32.0 (28.2) | 32.5 (28.2)

6. Primary Outcome: Birth Outcomes Head Circumference.
Description: Birth outcomes obtained from labor and delivery records head circumference measured in centimeters.
Time Frame: Postpartum
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 64 | 65
cm | 33.3 (1.7) | 33.0 (1.8)

7. Primary Outcome: Birth Outcomes 5-minute Appearance, Pulse, Grimace, Activity, and Respiration Score
Description: Birth outcomes obtained from labor and delivery records 5-minute Appearance, Pulse, Grimace, Activity, and Respiration score (APGAR). The Apgar score has a range from 0 to 10. A 5-minute Apgar score of 7-10 as reassuring, a score of 4-6 as moderately abnormal, and a score of 0-3 as low in the term infant and late-preterm infant 6.
Time Frame: postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 64 | 65
score on a scale | 8.9 (0.3) | 8.6 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time subjects received their first dose of study medication until the end of the 10-week treatment period or, if the adverse event was present at 10 weeks, until it resolved, up to 20 weeks.
Arm/Group | Placebo | Bupropion
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 3/65 | 2/64
Other Adverse Events (participants affected / at risk) | 40/65 | 41/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Bupropion (N=64)
Spontaneous delivery with Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Vasa previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth with Nuchal Cord (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Still birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Bupropion (N=64)
Nausea (General disorders) | 12 (15) | 11 (13)
Headache (Gastrointestinal disorders) | 10 (13) | 13 (16)
Vomiting (General disorders) | 9 (11) | 6 (7)
Constipation (General disorders) | 8 (8) | 6 (7)
Dry Mouth (Gastrointestinal disorders) | 7 (7) | 6 (10)
Irritability (Gastrointestinal disorders) | 6 (7) | 7 (11)
Sleep problem (Gastrointestinal disorders) | 9 (9) | 16 (18)
Fatigue (Gastrointestinal disorders) | 4 (4) | 4 (4)
Depressed Mood (General disorders) | 3 (3) | 4 (4)
Insomnia (Gastrointestinal disorders) | 3 (3) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02188459/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02188459/ICF_001.pdf